CLINICAL TRIAL: NCT02809573
Title: An Open-label, Multi-center, Phase Ib Clinical Trial of Chidamide Combined With CHOP in Newly Diagnosed Peripheral T-cell Lymphoma Patients
Brief Title: Clinical Trial of Chidamide Combined With CHOP in Peripheral T-cell Lymphoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDM103
Record Dates: First submitted 2016-06-17; First posted 2016-06-22 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: peripheral T-cell lymphoma; PTCL; chidamide; CHOP; phase Ib
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study drugs (Experimental): Lead-in period is 4 days. Patients take a single dose of Chidamide tablet, then off for 3 days before the first cycle begins. In the subsequent treatment cycles, Chidamide tablets are given orally on Day 1,4,8 and 11 of each cycle. Cyclophosphamide, adriacin and vincristine are given in intravenous infusion on Day 1. On Day 1 to 5, prednisone is given orally. Treatment cycles are repeated every 3 weeks .The combination therapy lasts for at most 6 cycles. Patients enter the single agent therapy if attained complete response after 6-cycle combination therapy. In this stage, patients take chidamide orally on Day 1, 4, 8 and 11 of each cycle.
  Interventions: Drug: Chidamide; Drug: cyclophosphamide; Drug: adriacin; Drug: vincristine; Drug: prednisone

INTERVENTIONS:
Drug: Chidamide — In the lead-in period, patients take a single dose of Chidamide tablet on the first day and then off for 3 days before the first cycle begins. In the subsequent treatment cycles, Chidamide tablets are given orally on Day 1,4,8 and 11 of each cycle.
  Other Names: CS055
Drug: cyclophosphamide — On Day 1, cyclophosphamide is given in a 20-minute intravenous (IV) infusion at 750 mg/m^2 in 5 minutes after chidamide administration
  Other Names: CTX
Drug: adriacin — On Day 1, Adriacin is given in a 20-minute IV infusion at 50 mg/m^2 soon after cyclophosphamide administration.
  Other Names: ADR
Drug: vincristine — On Day 1, vincristine is given in IV infusion at 1.4 mg/m^2 after adriacin administration.
  Other Names: VCR
Drug: prednisone — On Day 1 to 5, prednisone is given orally at 100 mg once a day
  Other Names: PED

SUMMARY:
The purpose of this dose-escalation study is to assess the safety and tolerability of treatment with Chidamide in a range of doses combined with CHOP in fixed dose in patients with newly diagnosed peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
The purpose of this study is to assess the tolerability and safety include adverse events, vital signs, laboratory tests, etc., of a range of doses of chidamide combined with CHOP in peripheral T-cell lymphoma patients, and to determine the dose limit toxicity and the maximum tolerable dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18-65 years old;
2. Histopathologically confirmed Peripheral T -cell Lymphoma (PTCL) including:

   * PTCL-unspecified;
   * Angioimmunoblastic T-cell lymphoma;
   * Anaplastic large cell lymphoma, ALK positive or negative;
   * Subcutaneous panniculitis T-cell lymphoma;
   * Cutaneous / T-cell lymphoma;
   * Other T-cell lymphoma that investigators consider to be appropriate to be enrolled;
3. Patients have not received anti-tumor therapy;
4. In any Ann Arbor disease stage;
5. ECOG performance status 0-1;
6. Patients without bone marrow involvement. The absolute number of neutrophile is no less then 2.0 * 10^9/L, platelet no less then 100 * 10^9/L. And the concentration of hemoglobin is no less than 110 g/L;
7. Life expectancy is no less than 6 months;
8. Patients who have signed the Informed Consent Form.

Exclusion Criteria:

1. Patients who have central nervous system or meninges involvements;
2. Patients have been treated by radiotherapy, chemotherapy or immunotherapy for PTCL;
3. Patients have uncontrollable or significant cardiovascular disease including:

   * history of myocardial infarction;
   * uncontrollable angina within the 6 months before screening, or taking anti-angina drugs at the time of screening;
   * history of congestive heart failure, or the left ventricular ejection fraction (LVEF) is < 50% at the time of screening;
   * clinically significant ventricular arrhythmia such as ventricular tachycardia, ventricular fibrillation or torsades de pointes;
   * History of supraventricular arrhythmia or nodal arrhythmia that could not been controlled by drug or need a pacemaker;
   * History of cardiomyopathy;
   * History of clinically significant QTc interval prolongation, or QTc interval > 450 ms at screening;
   * Coronary disease which is with symptoms and needs drug therapy;
4. Patients have undergone organ transplantation;
5. Patients with thromboembolic disease, hematencephalon or cerebral infraction within 4 weeks before screening, or patients who are under anticoagulant therapy;
6. Patients with clinically significant abnormalities in gastrointestinal tract, such as dysphagia, chronic diarrhea and intestinal obstruction which may affect the uptake,transformation and absorption of the drug;
7. Patients with active infections, including active bacterial,viral,fungoid, mycobacterium, parasite infections (but not including hyponychium fungoid infection), or infections which need not be treated by intravenous antibody therapies, or antiviral therapies, or any serious infection need to be treated by hospitalization;
8. Patients who have been conducted the surgery on a major organ in less than 6 weeks;
9. Hepatic function: Serum total bilirubin > 1.5 fold of normal range; ALT/AST > 2.5 folds of normal range or 5 folds for liver metastasis; Renal function: Serum creatine > 1.5 folds of normal range;
10. Patients with other malignancies in the past or now (except basal cell carcinoma, squamous-cell carcinoma or carcinoma in situs of cervix that has been adequately treated),unless the malignancy has been radically treated and there has been no evidence of recurrence for 5 years;
11. Pregnant or lactating women and patients in childbearing age who will not carry out birth control;
12. Patients with mental disorders, which may affect understanding and execution of informed consent or the compliance of the study;
13. Drug abuse or long term alcoholism that could affect the evaluation for the study results;
14. Patients considered by investigators not suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
dose-limiting toxicity (DLT) | Day 1 - 21

SECONDARY OUTCOMES:
Adverse events | About 21 weeks
complete response rate | About 21 weeks
Duration of response | About 21 weeks
Progression free survival | About 21 weeks
Objective response rate | About 21 weeks
Overall survival | About 21 weeks
Area under the concentration versus time curve (AUC) | Day 1 of the lead-in period and Day 1 of the combination therapy
Peak plasma concentration (Cmax) | Day 1 of the lead-in period and Day 1 of the combination therapy
Time of Cmax (Tmax) | Day 1 of the lead-in period and Day 1 of the combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided